CLINICAL TRIAL: NCT04208659
Title: Self-Administration of Auricular Acupuncture Pilot Project
Brief Title: Veteran Ear Acupuncture Pilot Project
Acronym: SAAAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chillicothe VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ChilliVASAAAUC2019-0194
Record Dates: First submitted 2019-12-12; First posted 2019-12-23 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain Syndrome; Pain; Fibromyalgia; Low Back Pain; Neuropathic Pain; Neuropathy, Painful; Musculoskeletal Pain; Chronic Pain
Keywords: acupuncture; auricular acupuncture; chronic pain; fibromyalgia; low back pain; lumbago; neuropathic pain; neuropathy; self-treatment; musculoskeletal pain; prosthesis-guided acupuncture; device-guided acupuncture; device-facilitated acupuncture
MeSH Terms: conditions — Pain; Fibromyalgia; Low Back Pain; Neuralgia; Neuropathy, Painful; Musculoskeletal Pain; Chronic Pain | interventions — Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: This is a pilot project to assess safety of self-administration of auricular acupuncture over a six-month period and how well a custom prosthesis facilitates needle placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-administration of Auricular Acupuncture Group (Experimental): There is only one arm in this pilot project, whose purpose is to determine safety of self-administration of Battlefield Acupuncture over a six month period and how well a prosthesis facilitates needle insertion. Five ASP (Aiguille D'acupuncture semi-permanente) needles will be self-inserted into each participant's ear every two weeks according to the standardized acupuncture points in Battlefield Acupuncture.
  Interventions: Procedure: Self-administration of auricular acupuncture without prosthesis; Procedure: Self-administration of auricular acupuncture with prosthesis

INTERVENTIONS:
Procedure: Self-administration of auricular acupuncture without prosthesis — Participants will insert semi-permanent acupuncture needles in their ears without the guidance of a prosthesis
Procedure: Self-administration of auricular acupuncture with prosthesis — The same participants who previous self-administered a standardized auricular acupuncture will be given custom-molded prostheses midway through the study to assess how much the prostheses facilitate insertion.

SUMMARY:
Veterans who have responded well to Battlefield Acupuncture (BFA), a form of auricular acupuncture, in routine clinical practice will be invited to receive education to insert the needles themselves at home. A 3D-printed wearable prosthetic will also be explored as a means to facilitate needle placement.

Primary end-points will include whether adverse events occur over a six-month period and whether the aforementioned prosthesis significantly facilitates needle placement in terms of subjective ease of administration.

DETAILED DESCRIPTION:
30 veterans who have repeatedly had good responses to BFA will be invited to participate. The PI and his collaborators will give standardized education (BFA training) to the veterans in a group session to teach them how to self-administer the BFA. The BFA training will be identical to that used by the VA for providers except that the training will focus on self-administration. The participants will be given needles in a manner similar to a prescription medication (i.e. controlled by the provider). They will self-administer BFA every two weeks for a total of 6 months and record their response in a standardized BFA template. Providers will call participants at intervals of two to four weeks to retrieve this data and assess for any adverse events other than minor bleeding, scratches and dizziness.

A plastic, custom-molded prosthesis will be developed during the first several months using 3D-scanning and 3D-printing. This prosthesis will be wearable over the ear and will have holes directly over the relevant acupuncture points to facilitate insertion. At the 3-month mark, participants will be given these. If this turns out to not be feasible with the available resources, work on this will cease for the remainder of the project. At the end of the study, participants will be asked whether the prosthesis made a significant difference in the ease of administration and open-ended comments regarding their experience will also be solicited.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic pain from any etiology
* Participant is physically and cognitively able to self-administer auricular acupuncture. This will be determined by the investigator during the educational sessions.
* Participants taking anti-coagulant or anti-platelet medications will be allowed to participate if they acknowledge an increased risk of bleeding

Exclusion Criteria:

* Condition causing ongoing immunocompromised state (e.g. overt AIDS, chemotherapy, anti-rejection medications)
* Acquired or congenital defects in the tympanic membrane
* Pregnancy
* Severe cognitive impairment
* Physical disability precluding self-administration of auricular acupuncture
* History of severe vasovagal reaction to acupuncture needling
* History of endocarditis
* History of artificial heart valve
* History of implanted device to support cardiac function
* Participation will be terminated for participants who use the acupuncture needles in any way other than instructed

Exclusion criteria include those who do not wish to participate and those who have significant contraindications to AA (auricular acupuncture) or indwelling acupuncture. These include: being immunocompromised, congenital or acquired defects in the tympanic membrane, pregnancy, severe cognitive impairment, inability to perform BFA on themselves. Medical anti-coagulation is not an automatic exclusion as many patients on these medications will not have any issues with bleeding with BFA. Those who have history of severe vasovagal/syncopal or other adverse response to skin puncture will also be excluded. Those with artificial heart valves or those with a history of heart valve infection are excluded because of risk of endocarditis. Pregnant patients will be excluded from this study to eliminate the possibility of harm to pregnant patients and developing children. Medical conditions that would exclude someone from using BFA include: 1) those with replacement heart valves; 2) those with history of heart valve infection; 3) those who are pregnant; 4) those who have a pacemaker, defibrillator, or other similar electronic device; 5) those who are afraid of needles, 6) those who are scheduled for an MRI; 7) those with non-medication induced bleeding disorders.

Participants will be removed from the study if it is discovered they are using the needles in a manner that is inconsistent with the protocol.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Self-Administered Auricular Acupuncture) | Six months
  The total number of self-reported adverse events other than minor self-limited bleeding (less than 1 mL per episode of acupuncture), dizziness and mild nausea will be recorded for the participants. The absolute number and percentage of participants experiencing adverse events greater than the aforementioned will be reported.
Incidence of Perceived Improved Ease of Self-administration of Auricular Acupuncture with 3D-printed Ear Prostheses | 3 months
  What percentage of patients affirm that the ear prostheses provided during the study make the self-administration of auricular acupuncture easier to perform? This is a dichotomous "yes/no" question.

SECONDARY OUTCOMES:
Comparative Satisfaction with Pain Control of Self-Administered Auricular Acupuncture versus Previous Episodes of Provider Administered Auricular Acupuncture | 6 months
  Previous provider-administered post-needling auricular acupuncture pain scores as measured by the Numeric Rating Scale will be averaged for each participant according to the availability of such data. All participants will be expected to have several such data points in the electronic medical record. These scores will be averaged for each patient. This individual average will be compared to the average of post-needling NRS scores reported from the self-administration of auricular acupuncture for the same patient. The percentage of difference in the NRS score between provider-administered and self-administered acupuncture will be reported to assess for possible non-inferiority of self-administered auricular acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Brian L James, MD, Principal Investigator — Chillicothe VA Medical Center
Locations (1):
- Chillicothe VA Medical Center, Chillicothe, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data from this small pilot project.

REFERENCES:
- [Background] White, A, Cummings, M, Filshie Jacqueline. An Introduction to Western Medical Acupuncture. Philadelphia, PA: Elsevier; 2008.
- [Background] Alimi D, MD, Geissmann A, MD, Gardeur D, MD. Auricular Acupuncture Stimulation Measured on Functional Magnetic Resonance Imaging, Medical Acupuncture. 2002:13(2);18-21.
- [Background] Goertz CM, Niemtzow R, Burns SM, Fritts MJ, Crawford CC, Jonas WB. Auricular acupuncture in the treatment of acute pain syndromes: A pilot study. Mil Med. 2006 Oct;171(10):1010-4. doi: 10.7205/milmed.171.10.1010. PMID 17076456
- [Background] Niemtzow RC, Burns SM, Cooper J, Libretto S, Walter JAG, Baxter J., Acupuncture Clinical Pain Trial in a Military Medical Center: Outcomes, Medical Acupuncture. 2008:20(4); 255-261
- [Background] Burns S, York A, Niemtzow RC, Garner BK, Steele N, Walter JAG. Moving Acupuncture to the Front Line of Military Medical Care; A Feasibility Study, Medical Acupuncture. 2013:25(1);48-54.
- [Background] Usichenko TI, Dinse M, Hermsen M, Witstruck T, Pavlovic D, Lehmann C. Auricular acupuncture for pain relief after total hip arthroplasty - a randomized controlled study. Pain. 2005 Apr;114(3):320-327. doi: 10.1016/j.pain.2004.08.021. PMID 15777857
- [Background] Vas J, Aranda-Regules JM, Modesto M, Aguilar I, Baron-Crespo M, Ramos-Monserrat M, Quevedo-Carrasco M, Rivas-Ruiz F. Auricular acupuncture for primary care treatment of low back pain and posterior pelvic pain in pregnancy: study protocol for a multicentre randomised placebo-controlled trial. Trials. 2014 Jul 16;15:288. doi: 10.1186/1745-6215-15-288. PMID 25027493
- [Background] Yeh CH, Chiang YC, Hoffman SL, Liang Z, Klem ML, Tam WW, Chien LC, Suen LK. Efficacy of auricular therapy for pain management: a systematic review and meta-analysis. Evid Based Complement Alternat Med. 2014;2014:934670. doi: 10.1155/2014/934670. Epub 2014 Jul 23. PMID 25165482
- [Background] Hou PW, Hsu HC, Lin YW, Tang NY, Cheng CY, Hsieh CL. The History, Mechanism, and Clinical Application of Auricular Therapy in Traditional Chinese Medicine. Evid Based Complement Alternat Med. 2015;2015:495684. doi: 10.1155/2015/495684. Epub 2015 Dec 28. PMID 26823672
- [Background] Chang LH, Hsu CH, Jong GP, Ho S, Tsay SL, Lin KC. Auricular acupressure for managing postoperative pain and knee motion in patients with total knee replacement: a randomized sham control study. Evid Based Complement Alternat Med. 2012;2012:528452. doi: 10.1155/2012/528452. Epub 2012 Jul 10. PMID 22844334
- [Background] Fox LM, Murakami M, Danesh H, Manini AF. Battlefield acupuncture to treat low back pain in the emergency department. Am J Emerg Med. 2018 Jun;36(6):1045-1048. doi: 10.1016/j.ajem.2018.02.038. Epub 2018 Feb 27. PMID 29550099
- [Background] Jan AL, Aldridge ES, Rogers IR, Visser EJ, Bulsara MK, Niemtzow RC. Does Ear Acupuncture Have a Role for Pain Relief in the Emergency Setting? A Systematic Review and Meta-Analysis. Med Acupunct. 2017 Oct 1;29(5):276-289. doi: 10.1089/acu.2017.1237. PMID 29067138
- [Background] Lee RJ, McIlwain JC. Subacute bacterial endocarditis following ear acupuncture. Int J Cardiol. 1985 Jan;7(1):62-3. doi: 10.1016/0167-5273(85)90175-5. PMID 4055136
- [Background] Stellon A. Acupuncture in patients with valvular heart disease and prosthetic valves. Acupunct Med. 2003 Sep;21(3):87-91. doi: 10.1136/aim.21.3.87. PMID 14620303
- [Background] Tan JY, Molassiotis A, Wang T, Suen LK. Adverse events of auricular therapy: a systematic review. Evid Based Complement Alternat Med. 2014;2014:506758. doi: 10.1155/2014/506758. Epub 2014 Nov 10. PMID 25435890
- [Derived] James BL, Welch J, Williamson C. Self-Administration of Auricular Acupuncture in Rural Veterans with Chronic Pain: A Pilot Project. Med Acupunct. 2021 Oct 1;33(5):349-352. doi: 10.1089/acu.2021.0007. Epub 2021 Oct 18. PMID 35003503

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04208659/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04208659/ICF_000.pdf